CLINICAL TRIAL: NCT01714570
Title: A Prospective, Randomized, Open Label Study of Piperacillin/Tazobactam Versus Imipenem/Cilastin for Empirical Therapy of Febrile Patients With Neutropenia After Hematopoietic Stem Cell Transplantation
Brief Title: Piperacillin/Tazobactam for Empirical Therapy of Febrile Neutropenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Wenrong Huang, Associate director, Hematology, Chinese PLA General hospital, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTZ-20120702
Record Dates: First submitted 2012-07-04; First posted 2012-10-26 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Febrile; Neutropenia; Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Fever; Neutropenia | interventions — Piperacillin, Tazobactam Drug Combination; Imipenem; Cilastatin, Imipenem Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- piperacillin/tazobactam (Experimental)
  Interventions: Drug: Piperacillin-tazobactam combination product
- imipenem/cilastatin (Active Comparator)
  Interventions: Drug: Imipenem

INTERVENTIONS:
Drug: Piperacillin-tazobactam combination product — 4.5g q6h, 5-10 days
  Other Names: Tazocin
  Arms: piperacillin/tazobactam
Drug: Imipenem — 0.5g q6h, 5-10 days
  Other Names: Tienam
  Arms: imipenem/cilastatin

SUMMARY:
Neutropenia is very common in patients received hematopoietic stem cell transplantation, with median duration of about 14 days. In 2010 update, IDSA recommended Piperacillin/tazobactam as first-line mono-therapy for febrile patients with neutropenia of high risk. In china, the data of piperacillin/tazobactam for febrile neutropenia after hematopoietic stem cell transplantation is very limited.

The current study will evaluate the efficacy of piperacillin/tazobactam compared with imipenem/cilastatin for febrile neutropenia after transplantation.

DETAILED DESCRIPTION:
1. Swab culture (skin, pharyngeal, nasal, anus) when administered into laminar flow room after transplantation.
2. Randomize the febrile patients into 2 groups.
3. Therapy group receive piperacillin/tazobactam, 4.5g q6h iv. Control group receive imipenem/cilastatin, 0.5g q6h. Duration will be 5-10 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-65 years
* received Autologous or Allogeneic hematopoietic stem cell transplantation.
* ECOG score 0-1.
* ICF is available.

Exclusion Criteria:

* Allergic to any therapy drug.
* Documented infection before neutropenia.
* Renal dysfunction.
* Suffering from central nervous system or mental disease.

Ages: 13 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Clinical success rate. | 3 weeks after beginning of empirical therapy
  Resolve of clinical symptoms and signs, without change of therapy.

SECONDARY OUTCOMES:
Microbiologic success rate | 3 weeks after beginning of empirical therapy
  Microbiologic success includes eradication, suspected eradication, and super-infection.
  1. Eradication or Presumed eradication: the baseline pathogens no longer present on the culture performed after completion of treatment. If no way to collect biologic sample(s) after treatment;, e.g. sputum, a presumed eradication will be concluded
  2. No eradication: one or more baseline pathogens were persistent
  3. Relapse: the baseline pathogens transient absence reappeared during the therapy
  4. Alternative: the baseline pathogens were eradicated, but new ones appeared without any clinical signs and symptoms
  5. Re-infection: the baseline pathogens were eradicated, but new ones appeared with clinical signs and symptoms.
Adverse effect | 3 weeks after beginning of empirical therapy
  The number of patients developed unexpected medical information at the 3 weeks after beginning of empirical therapy.
Cost of drug and therapy | 3 weeks after beginning of empirical therapy

CONTACTS AND LOCATIONS:
Overall Officials: wenrong huang, Doctor, Principal Investigator — Employee
Locations (1):
- Chinese PLA general hospital, Beijing, Beijing Municipality, China